CLINICAL TRIAL: NCT05898321
Title: A Multicenter，Prospective Clinical Trial for Reducing Remaining Submucous Fibroids Volume and Preventing Recurrence by Treating With GnRH Analogues or Mifepristone After Transcervical Resection of Type I-II Myoma
Brief Title: To Prevent Type I-II Myoma After TCRM Recurrence by Gonadotropin-releasing Hormone (GnRH )Analogues or Mifepristone
Acronym: TCRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-20230046-R
Record Dates: First submitted 2023-02-10; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Submucous Leiomyoma of Uterus
Keywords: Submucous leiomyoma; Transcervical resection of myoma; GnRH analogues
MeSH Terms: interventions — Goserelin; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GnRHa group (Experimental): Patients with fibroid remained will be enrolled and one third of them will be administrated with Zoladex (3.60mg/28 days) for three to six months,.
  Interventions: Drug: Zoladex
- mifepristone group (Experimental): Patients with fibroid remained will be enrolled and one third of them will be administrated with mifepristone(10.0mg/d) for three to six months.
  Interventions: Drug: Mifepristone Oral Tablet
- control group (No Intervention): Patients with fibroid remained will be enrolled and the third group was serviced as controls and no drugs will be used.

INTERVENTIONS:
Drug: Zoladex — Patients with fibroid remained will be enrolled and divided into three groups. one group wii be administrated with Zoladex (3.60mg/28 days) for three to six months.
  Arms: GnRHa group
Drug: Mifepristone Oral Tablet — Patients with fibroid remained will be enrolled and divided into three groups. one group will be administrated with mifepristone(10.0mg/d) for three to six months.
  Arms: mifepristone group

SUMMARY:
Transcervical resection of myoma(TCRM) has a good therapeutic effect while the probability of complete resection of type I and II fibroids is only 55% per procedure on average and a significant number of patients have fibroid remained.At present, there is no standardized treatment option for reducing the remaining submucous fibroids volume and preventing its recurrence after TCRM.The present prospective,multicentre,randomised controlled clinical trial will enrol women after TCRM and treat them with mifepristone(10mg)or GnRHa(3.60mg)for 3 to 6 months,investigating the effective and cost-effective treatment options after fibroids with TCRM，thus to provide evidence and effectual regiments for reducing remaining fibroids volume and preventing its recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years and less than 45 years old, no childbirth requirements in the next 3 years;
2. Type I and II submucosal fibroids diagnosed by ultrasound, and the diameter of them are greater than 3cm;
3. Type I or II submucosal fibroids confirmed by TCRM and no degeneration confirmed pathologically;
4. A MRI test will be done to evaluate the residual submucosal fibroids and calculate the residual fibroid volume after 1 month of surgery;
5. Patients would not had used drugs such as mifepristone and GnRHa 3 months before surgery;
6. Participate in this trial and sign the informed consent form voluntarily .

Exclusion Criteria:

1. Combined with congenital uterine malformations such as double uterus, unicornuate uterus, etc;
2. Have fertility requirements within 3 years after surgery;
3. Estrogen-dependent diseases such as adenomyosis and endometriosis;
4. Drugs such as mifepristone or GnRHa have been used before surgery;
5. Mifepristone or GnRHa drug treatment is contraindicated or cannot tolerate TCRM surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 294 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the remaining submucous fibroids volume | one to three years after TCRM
  The change of residual fibroid volume is compared to residual fibroid volume measured by ultrasound and /or MRI one month after surgery;

SECONDARY OUTCOMES:
the recurrence rate of remaining submucous fibroids and time | one to three years after TCRM
  recurrent submucosal fibroids include increased menstrual flow and continued growth of residual submucosal fibroids.
the recurrence time of remaining submucous fibroids | one to three years after TCRM
  the time interval between recurrent submucosal fibroids and TCRM

CONTACTS AND LOCATIONS:
Overall Officials: Lv weiguo, Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No